CLINICAL TRIAL: NCT01223976
Title: Sensitivity and Specificity of QuantiFeron -TB Gold Test (QFT-G)in Comparison With Tuberculin Skin Test in Patients With Psoriasis and Psoriatic Arthritis
Brief Title: Sensitivity and Specificity of QuantiFeron -TB Gold Test (QFT-G)in Patients With Psoriasis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof. Ori Elkayam, Tel Aviv Medical Center
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 222-10
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Tuberculosis; Psoriasis
Keywords: latent tuberculosis psoriasis arthritis TST QTF; Screening of latent tuberculosis in psoriasis
MeSH Terms: conditions — Tuberculosis; Psoriasis | interventions — Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Tuberculin skin test and Quantiferon -TB Gold test — TST A 2-TU dose of PPD will bevadministered by a certified technician using the Mantoux method and induration measured after 72 h.
  QFT-G test The second-generation QuantiFeron® (QIFN) whole-blood IFN assay (Cellestis) will be performed and interpreted according to the manufacturer's instructions.

SUMMARY:
The purpose of this study is to determine the level of agreement between QuantiFeron -TB Gold test (QFT-G)and Tubeculin skin test (TST)for screening of latent tuberculosis in patients suffering from psoriasis.

DETAILED DESCRIPTION:
Patients with psoriasis and psoriatic arthritis are candidates to receive anti-TNF alpha therapies which require prior screening for latent tuberculosis (LTB). Currently, screening for LTB is based on tuberculin skin test (TST) , chest X rays, and a questionaire on predisposing factors for TB. The main drawbacks of TST are the lack of specificity due to cross reactivity with Bacille Calmette- Guerin (BCG) and other nontuberculosis mycobacteria and the risk of anergy in immunosuppressed patients. Furthermore, it has been suggested that the skin of psoriatic patients may be more sensitive resulting in increased TST which does not obligatory reflect the status of LTB.

Recently, a new assay for LTBI has been developed, which evaluates interferon (IFN) -γ release by memory effector T-cells stimulated in vitro with specific mycobacterial antigens, ESAT-6 (early secretory antigen target-6) and CFP-10 (culture filtrate protein-10) [9-10]. The QuantiFeron -TB Gold test (QFT-G) uses ELISA to measure IFN-γ concentrations in supernatants in plate format and "In tube" format (QFT-GIT) while the enzyme-linked immunospot (ELISPOT) detects individual IFN-γ producing T-cells (TS-TB, Oxford Immunotech, Abingdon, UK).

The whole blood IFN-γ assays was approved by The Centers for Disease Control as an alternative screening strategy to TST in immunocompetent individuals [11], but its clinical utility as a single test for detection LTBI in immunocompromised patients is controversial.Furthermore, its utility in patients with psoriasis and psoriatic arthritis has not been yet established One hundred patients with psoriasis and psoriatic arthritis and 50 healthy control will participate in this study.

Enrolled subjects will be requested to complete a detailed sociodemographic and TB screening questionnaire including gender, age, place of birth and work, prior BCG vaccination, close contact with TB patients or TB prophylaxis in the past. Screening workup will includ assessment of clinical disease activity using the Disease Activity Score 28 (DAS-28)and Psoriasis Area Severity Index (PASI),documentation of past or current treatment with systemic corticosteroids and immunosuppressive drugs, and imaging (chest X-ray).

All the subjects will undergo a TST and QFT-G test A 2-TU dose of PPD will be administered by a certified technician using the Mantoux method and induration measured after 72 h. TST will be deemed positive if bove or equally to 5 mm for RA patients and 10 mm for controls The absence of induration of <2 mm in diameter will be recorded as anergic and negative TST results was defined as having more than 2 but less than 5 mm reactions for RA patients.

QFT-G test The second-generation QuantiFeron® (QIFN) whole-blood IFN assay (Cellestis) will be performed and interpreted according to the manufacturer's instructions.

Briefly, the test consisted of a negative control (nil well, i.e., whole blood without antigens or mitogen),a positive control (mitogen well, i.e., whole blood stimulated with the mitogen phytohemagglutinin [PHA]) and two sample wells, i.e., whole blood stimulated with either of the M. tuberculosis-specific antigens, Early Secretory Antigen Target 6 (ESAT-6) or Culture Filtrate Protein 10 (CFP-10).

Five ml heparinized whole blood will be drawn for QFT-G before for PPD testing. The blood specimens will be incubated for 16-20 h (overnight) at 37°C in a humidified atmosphere. IFN-γ levels in the nil well will be considered background and will be subtracted from the results of the mitogen well and the antigen-stimulated wells. The results will be considered positive if the concentration of.IFN-γ in the sample well after stimulation with ESAT-6 and/or CFP-10 will be greater than or equal to 0.35 IU/ml (after subtracting the value of the nil well), regardless of the results of the positive control (mitogen well). The results will be considered negative if the response to the specific antigens (after subtracting the value of the nil well) is less than 0.35 IU/ml and if the IFN-γ levels of the positive control (after subtracting the value of the nil well) is greater than or equal to 0.5 IU/ml. The results will be considered indeterminate if both antigen-stimulated sample wells are negative (i.e., <0.35 IU/ml after subtracting the value of the Nil well) and if the value of the positive control well is less than 0.5 IU/ml after subtracting the value of the nil well

the nil well.

QFT-G test The second-generation QuantiFeron® (QIFN) whole-blood IFN assay (Cellestis) was performed and interpreted according to the manufacturer's instructions.

Briefly, the test consisted of a negative control (nil well, i.e., whole blood without antigens or mitogen) , a positive control (mitogen well, i.e., whole blood stimulated with the mitogen phytohemagglutinin [PHA]) and two sample wells, i.e., whole blood stimulated with either of the M. tuberculosis-specific antigens, Early Secretory Antigen Target 6 (ESAT-6) or Culture Filtrate Protein 10 (CFP-10).

Five ml heparinized whole blood was drawn for QFT-G before for PPD testing. The blood specimens were incubated for 16-20 h (overnight) at 37°C in a humidified atmosphere. IFN-γ levels in the nil well were considered background and were subtracted from the results of the mitogen well and the antigen-stimulated wells. The results were considered positive if the concentration of. IFN-γ in the sample well after stimulation with ESAT-6 and/or CFP-10 was greater than or equal to 0.35 IU/ml (after subtracting the value of the nil well), regardless of the results of the positive control (mitogen well). The results were considered negative if the response to the specific antigens (after subtracting the value of the nil well) was less than 0.35 IU/ml and if the IFN-γ levels of the positive control (after subtracting the value of the nil well) were greater than or equal to 0.5 IU/ml. The results were considered indeterminate if both antigen-stimulated sample wells were negative (i.e., <0.35 IU/ml after subtracting the value of the Nil well) and if the value of the positive control well was less than 0.5 IU/ml after subtracting the value of

the nil well.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis and psoriatic arthritis
* Aged 18-90

Exclusion Criteria:

* History of TB
* Known allergy to TST
* Current or past treatment with anti-TNF alpha

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
The level of agreement between TST and QTF in patients with psoriasis in comparison with controls | 3 days

SECONDARY OUTCOMES:
Levels of TST in patients with psoriasis in comparison with healthy controls | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Chiang YZ, Panting K, Dever B, Parslew RA. Clinical applicability of T-cell interferon-a release assay for tumour necrosis factor-a inhibitor therapy in severe psoriasis. Clin Exp Dermatol. 2011 Jan;36(1):39-41. doi: 10.1111/j.1365-2230.2010.03850.x. PMID 20456401
- [Background] Laffitte E, Janssens JP, Roux-Lombard P, Thielen AM, Barde C, Marazza G, Panizzon RG, Saurat JH. Tuberculosis screening in patients with psoriasis before antitumour necrosis factor therapy: comparison of an interferon-gamma release assay vs. tuberculin skin test. Br J Dermatol. 2009 Oct;161(4):797-800. doi: 10.1111/j.1365-2133.2009.09331.x. Epub 2009 Jun 5. PMID 19659473